CLINICAL TRIAL: NCT01054976
Title: The Efficacy of Galantamine Treatment on Attention in Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015850; GAL-KOR-21 (Other: Janssen Korea, Ltd., Korea); GALALZ4039 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Results first posted 2012-12-24 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-11

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; Galantamine; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Galantamine

ARMS (1):
- Galantamine (Experimental)
  Interventions: Drug: Galantamine

INTERVENTIONS:
Drug: Galantamine — Orally administered Galantamine 8 mg/day for the first 4 weeks. Thereafter the dose will be increased to 16 mg/day. If tolerated, the dose of galantamine can be increased up to 24 mg/day.

SUMMARY:
This study will examine whether the administration of galantamine is effective for improvement of attention and more effective for patients with serious disturbance of attention by administering galantamine to patients with Alzheimer's dementia and performing an attention test on baseline, week 4 and 12.

DETAILED DESCRIPTION:
This is an open label (all people know the identity of the intervention), multi-center, prospective study investigating the effect of galantamine on the attention of Alzheimer's dementia patients. The objectives of this study include the evaluation of the relationship between change in attention after 4 weeks of galantamine administration and to investigate the effect of study drug after 12 weeks administration (the difference in the improvement of attention after the administration of galantamine). The secondary objective of this study is to clarify the causal relationship between improvement of attention and activities of daily living (ADL). The design of this study is prospective, open-label, multi-center study. Study populations are probable Alzheimer's dementia patients diagnosed by NINCDS-ADRDA (National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's disease and Related Disorders Association), DSM-IV (Diagnostic and Statistical Manual of Mental Disorders) criteria. The efficacy of study drug will be assessed by evaluating cognitive function, attention and behavioral symptoms before and after the treatment using the following assessment tools: ADAS-K-cog11 (Alzheimer's Disease Assessment Scale - cognitive subscale), computerized attention test and activities of daily living. Safety evaluations include adverse event monitoring and clinical lab tests. The patient is administered oral galantamine 8 mg/day for the first 4 weeks and then 16 mg/day. The dose of galantamine is increased up to 24 mg if tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's disease according to the criteria of DSM-IV, NINCDS-ADRDA
* K-MMSE (Korean - Mini Mental State Exam) is 10 to 24
* Reliable Guardian available to the patients
* Patient or guardian provided written informed consent before entering into the clinical trial

Exclusion Criteria:

* Acetylcholine esterase inhibitors used to treat dementia taken within 30 days of the beginning in this clinical trial
* Neurodegenerative diseases (eg Parkinson's disease, Pick's disease, Huntington's disease, Down syndrome)
* Dementia related to head trauma and dementia related to brain damage due to cerebral hypoxia (hypoxic brain damage after cardiopulmonary resuscitation, hypoxic brain damage after surgery, hypoxic brain damage due to addiction, hypoxic brain damage due to shock)
* brain tumor, nerve syphilis, meningitis, encephalitis
* epilepsy

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2006-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the total of 99 enrolled patients, only 92 were screened.
Groups:
- Galantamine: 8 mg/day for 4 weeks; 16 mg/day thereafter
Period: Overall Study
Arm/Group | Galantamine
Started | 92
Completed | 57
Not Completed | 35
Not completed — Adverse Event | 16
Not completed — Uncooperative participations to study | 7
Not completed — Withdrawal by Subject | 4
Not completed — Other | 8

BASELINE CHARACTERISTICS:
Arm/Group | Galantamine
Number analyzed (Participants) | 92
Age Continuous [Mean (Standard Deviation); unit: Years] | 73.24 (7.969)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Simple Reaction Time
Description: The Simple Reaction Time is a computerized attention test that evaluates the patient's reaction time when the color of the computer screen changes from black to white by performing a total of 70 times for six minutes.
Time Frame: Baseline, Week 12
Population: Per-protocol (PP) analysis set.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Galantamine
Number analyzed (Participants) | 92
seconds
  Week 4 (n=83) | -30.92 (1277.0)
  Week 12 (n=73) | 180.83 (519.18)

2. Primary Outcome: Change From Baseline in Choice Reaction Time
Description: The Choice Reaction Time is a computerized attention test that evaluates the reaction time and the number of errors by showing patients one card on the computer screen and making them find the same one among similar four cards. The test is performed a total of 12 times.
Time Frame: Baseline, Week 12
Population: Per-protocol (PP) analysis set.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Galantamine
Number analyzed (Participants) | 92
seconds
  Week 4 (n=80) | 429.54 (3388.0)
  Week 12 (n=73) | 1331 (3627.0)

3. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog)
Description: The Alzheimer's disease Assessment Scale-Cognitive subscale (ADAS-Cog) is an instrument used to assess cognitive dysfunction in individuals with Alzheimer disease and other dementias. It consists of 11 items, with scores ranging from 1 to 70. Maximum score is 70. Higher scores indicate worsening.
Time Frame: Baseline, Week 12
Population: Intention-to-Treat analysis set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Galantamine
Number analyzed (Participants) | 73
scores on a scale | 1.31 (5.67)

4. Secondary Outcome: Change From Baseline in Korean Version of Disability Assessment for Demential Scale (DAD-K)
Description: DAD-K is the Korean version of the Assessment for Dementia Scale, a tool developed to evaluate the Alzheimer patients' function including both basic and instrumental Activities of Daily Livings (ADL). It evaluates one function from various perspectives including behavior initiation, plan and preparation, and valid performance. It consists of 10 questions, each can score either 0 (no) or 1 (yes), if not applicable, patient will check on "not applicable (x)" which will not count in the calculation. Scores range from 0 to 100. Higher score represents better function
Time Frame: Baseline, Week 12
Population: Intention-to-Treat analysis set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Galantamine
Number analyzed (Participants) | 73
scores on a scale | -1.41 (10.53)

5. Secondary Outcome: Change From Baseline in Seoul-Instrumental Activities of Daily Livings (S-IADL)
Description: The Seoul-Instrumental Activities of Daily Living (S-IADL) assesses patients' abilities to perform instrumental and social activities of daily living. These include the ability to prepare a balanced meal, remember appointments, keep financial records, remember to take medication, and so on. It is composed of 15 items, with scores ranging from 0 to 45. Lower scores indicate better functioning.
Time Frame: Baseline, Week 12
Population: Intention-to-Treat analysis set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Galantamine
Number analyzed (Participants) | 73
scores on a scale | 1.22 (6.88)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Galantamine
Serious Adverse Events (participants affected / at risk) | 8/92
Other Adverse Events (participants affected / at risk) | 41/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Galantamine (N=92)
Fall (Injury, poisoning and procedural complications) | 2
Fracture (Injury, poisoning and procedural complications) | 2
Asthenia (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Headache (General disorders) | 1
Delirium (Psychiatric disorders) | 1
Brain stem infarction (Nervous system disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Neuromyopathy (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Galantamine (N=92)
Nausea (Gastrointestinal disorders) | 15
Dizziness/vertigo (Nervous system disorders) | 7
Anorexia (Nervous system disorders) | 6
Headache (General disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 4
Chest discomfort (Cardiac disorders) | 2
Weight loss (Metabolism and nutrition disorders) | 2
Insomnia (General disorders) | 2
Poor appetite (Metabolism and nutrition disorders) | 2
Asthenia (Musculoskeletal and connective tissue disorders) | 2
Cold (General disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Lethargy (General disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 2
Fall (General disorders) | 1
Fatigue (General disorders) | 1
Belching (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Sleep disorder (General disorders) | 1
Depression (Psychiatric disorders) | 1
Dementia (Psychiatric disorders) | 1
Sun stroke (General disorders) | 1
Tonic pain (Nervous system disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Hearing loss (Ear and labyrinth disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Rigor (Musculoskeletal and connective tissue disorders) | 1
Sweating (General disorders) | 1
Knee pain (Musculoskeletal and connective tissue disorders) | 1
Somnolence (General disorders) | 1
Confusion (Psychiatric disorders) | 1
Intermittent indigestion (Gastrointestinal disorders) | 1
Tremor (Nervous system disorders) | 1

LIMITATIONS AND CAVEATS:
A relatively low number of patients finished the study, which may have had an impact on the statistical power of data analysis. Difficulties in performing computer-based tests for elderly patients may have hampered detection of changes in attention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release (time limit not indicated).